CLINICAL TRIAL: NCT06002399
Title: Combining a Monofocal With an EDOF IOL: Is There an Improvement in Quality of Vision After Cataract Surgery Over Bilateral Monofocal IOL Implantation.
Brief Title: Bilateral Monofocal Versus Monofocal-EDOF IOL Implantation: Quality of Vision Comparison
Acronym: COMEDI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Karolien Termote, MD FEBOpht, Clinical Staff Member Ophthalmology, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23219_EDOF study
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral monofocal intraocular lens (Other): Standard treatment
  Interventions: Device: cataract surgery
- Monofocal and contralateral extended depth-of-focus intraocular lens (Experimental): Experimental treatment
  Interventions: Device: cataract surgery

INTERVENTIONS:
Device: cataract surgery — cataract surgery

SUMMARY:
The goal of this clinical trial is to compare visual quality after cataract surgery between two groups: bilateral monofocal intraocular lenses (IOL) and monofocal and contralateral extended depth-of-focus (EDOF) IOL implantation. The main question it aims to answer is:

• does the combination of both monofocal and EDOF IOLs presents an advantage over bilateral monofocal IOL implantation in the daily life of patients undergoing cataract surgery without the disadvantages of bilateral EDOF IOL implantation?

Participants will:

* be randomised in either bilateral monofocal group or monofocal and EDOF group
* undergo visual acuity testing with and without correction at all distances
* be asked to complete a quality of vision questionnaire
* undergo non-invasive examinations to measure residual astigmatism, contrast sensitivity, straylight, optical aberrations, reading spead.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 50 and 90 years with bilateral cataract without concomitant exclusion criteria

Exclusion Criteria:

* prior refractive surgery
* patients with corneal opacities, retinopathy, opticopathy, glaucoma, uveitis and amblyopia
* patients with corneal astigmatism greater than 3 diopters (D)
* patients with expected postoperative astigmatism higher than 0.50D
* prior ocular surgery in the last six months
* patients with prior unilateral cataract surgery

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Difference in binocular photopic distance corrected intermediate visual acuity between both groups using Radner chart. | 3 months
  Difference in binocular photopic distance corrected intermediate visual acuity between both groups using Radner chart.

REFERENCES:
- [Derived] Termote K, Van Schoor R, Krolo I, Oellerich S, Cools W, Delbeke H, Ni Dhubhghaill S. Combination of a monofocal and one type of extended depth-of-focus (zonal refractive) intraocular lens (COMEDI) in bilateral cataract surgery protocol: a monocentric, randomised, parallel group trial in cataract surgery. BMJ Open Ophthalmol. 2024 Aug 5;9(1):e001572. doi: 10.1136/bmjophth-2023-001572. PMID 39103234